CLINICAL TRIAL: NCT03158441
Title: DTi Diffusion Findings in Breast MRI Screening and Diagnostic
Status: Withdrawn | Type: Observational
Why Stopped: for technical and funding issues
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Ahuva Grubstein, head of mammography, Rabin Medical Center
Other Study IDs: 0425-16-RMC
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: MRI; Diffusion; DTI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: The patients enrolled for the study will be women scheduled for breast MRI due to high risk screening or pretreatment evaluation. The patients will fill in a form regarding: age, hormonal status, risk factors, prior breast surgery or treatment (a form which is routinely filled out in our institution). They will then undergo a breast MRI scan, using the routine protocol in our institution. This will be directly followed by a DTI sequence, which takes about 10 minutes in addition to the regular examination. The DTI sequence is routinely used in other imaging institutions, as part of the breast MRI protocol.
  Interventions: Diagnostic Test: Breast MRI
- control: same patients , dynamic scan
  Interventions: Diagnostic Test: Breast MRI

INTERVENTIONS:
Diagnostic Test: Breast MRI — comparison of DTI to dynamic MRI

SUMMARY:
Introduction The most common breast cancer originates within the breast milk ducts, and is called ductal carcinoma. After the stage where the cancer is found only within the ducts, it invades the breast tissue beyond the ducts, and becomes invasive cancer (Infiltrating Duct Carcinoma). Breast cancer located within the ducts is called intra ductal carcinoma in situ- DCIS. DCIS is the developing cancer and usually does not metastasize. Another type of breast cancer originates within the breast lobules and is call lobular carcinoma.

Recently at the Weizmann Institute, Prof. Hadassa Degani and her group developed and imaging technique using breast MRI. This technique allows to map the three-dimensional structure of the milk ducts in the breast. The method is based on measuring the random movement (Brownian motion) of water molecules (diffusion) in different directions in the breast tissue, collecting diffusion images by using magnetic field gradients in different directions, allowing imaging of Diffusion tensor Imaging -DTI. Movement of water molecules within a unified solution is usually random and uniform in all directions, but the internal structures in biological systems (such as cells, pipelines, fiber) restrict the movement of water in certain directions. The DTI method exploits this feature by measuring the diffusion in various directions, thus enabling calculating images of biological structures [1]. This method was proved to be effective in mapping the brain's white matter fibers and is used routinely in clinical tests used to monitor neurological injuries [2-4]. This method was used for milk ducts mapping within breast tissue at the Weizmann Institute. The system that was developed at the Weizmann Institute, showed that the movement of water molecules along the milk ducts is faster than their movement across the ducts and therefore it was possible using this method to map the breast ductal system. Also this method showed that it is possible to detect and diagnose malignant changes within breast and to distinguish them from normal tissue and benign tumors using DTI. Changes in cell density and arrangement causes changes in the directional diffusion coefficients and the differences between them [5-9] Research Plan Summary A prospective preliminary study to evaluate the correlation between the DTI analysis of breast MRI and the results of conventional contrast enhanced breast MRI.

The patients enrolled for the study will be women scheduled for breast MRI due to high risk screening or pretreatment evaluation. The patients will fill in a form regarding: age, hormonal status, risk factors, prior breast surgery or treatment (a form which is routinely filled out in our institution). They will then undergo a breast MRI scan, using the routine protocol in our institution. This will be directly followed by a DTI sequence, which takes about 10 minutes in addition to the regular examination. The DTI sequence is routinely used in other imaging institutions, as part of the breast MRI protocol.

The exams will be read on our regular work stations, and in addition will be analyzed by software developed at the Weizmann Institute. Both interpretations will then be compared to each other and to clinical and pathological data

ELIGIBILITY:
Inclusion Criteria:

- all patients undergoing breast MRI

Exclusion Criteria:

general contraindication to MRI -

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The patients enrolled for the study will be women scheduled for breast MRI due to high risk screening or pretreatment evaluation. The patients will fill in a form regarding: age, hormonal status, risk factors, prior breast surgery or treatment (a form which is routinely filled out in our institution). They will then undergo a breast MRI scan, using the routine protocol in our institution. This will be directly followed by a DTI sequence, which takes about 10 minutes in addition to the regular examination. The DTI sequence is routinely used in other imaging institutions, as part of the breast MRI protocol.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
DTI results as compre to dynamic scan results | 1 year
  colored scaling of DTI ranging from green to yellow and red as compare dynamic scan

CONTACTS AND LOCATIONS:
Overall Officials: Ahuva Grubstein, MD, Principal Investigator — Tel Aviv University

IPD SHARING:
Plan to Share IPD: Undecided